CLINICAL TRIAL: NCT02577146
Title: The Predictive Value of Ureteral Jet Assessment With Ultrasound in Patients Presenting With Acute Renal Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Midwest Stone Institute. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201506127
Record Dates: First submitted 2015-09-29; First posted 2015-10-16 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Ureteral Calculi
Keywords: stone; ureter; ultrasound
MeSH Terms: conditions — Ureteral Calculi; Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study ultrasound (Experimental): Study ultrasound with ureteral jet assessment will be obtained after CT diagnosis of ureteral calculus is made. Ureteral jet data will be documented and patients will be followed prospectively for 42 days for spontaneous stone passage or need for surgical intervention.
  Interventions: Device: renal and bladder ultrasound with ureteral jet assessment

INTERVENTIONS:
Device: renal and bladder ultrasound with ureteral jet assessment — The number of jets from each ureteral orifice will be tabulated over time so that ureteral jet frequency, defined as number of jets per minute, can be calculated. Patients will be categorized into three groups. Group I- no ureteral jets on the symptomatic side; Group II- continuous low-level ureteral jet on the symptomatic side; Group III- ureteral jets similar to nonsymptomatic side.

SUMMARY:
This is a single institution, prospective study to evaluate the prognostic significance of renal and bladder ultrasound with ureteral jet assessment and its utility to evaluate the spontaneous stone passage rate of ureteral stones.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older at the time of consent
* willing and able to sign consent
* CT diagnosis of ureteral stone with a stone burden less than or equal to 10mm

Exclusion Criteria:

* obstructed solitary kidney
* obstructed transplant kidney
* bilateral obstructed kidneys
* any condition or reason that, in the opinion of the treating physician, interferes with the patient's ability to participate or places the patient at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-10; Primary Completion 2018-05-07 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alana Desai, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Ultrasound
Started | 74
Completed | 46
Not Completed | 28
Not completed — Lost to Follow-up | 8
Not completed — Physician Decision | 3
Not completed — Screen Failure | 17

BASELINE CHARACTERISTICS:
Arm/Group | Study Ultrasound
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Time in Days From Diagnosis to Stone Passage.
Description: Number of days that have elapsed from date of diagnosis to date of stone passage or intervention to maximum observation time (42 days).
Time Frame: 42 days
Population: 28 cases were not included in analysis due to screen failures, subject non-compliance and missing data.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Study Ultrasound
Number analyzed (Participants) | 46
Days
  Present Jets: number analyzed (Participants) | 31
  Present Jets | 5 [3 to 13]
  Absent Jets: number analyzed (Participants) | 15
  Absent Jets | 13 [8 to NA] — Sample size is too small to estimate upper limit of 95% confidence interval.

2. Secondary Outcome: The Number of Cases With Concordant Treatment Recommendations Based on the Ultrasound and CT Scan.
Time Frame: 42 days
Population: 28 cases were not included in analysis due to screen failures, subject non-compliance and missing data.
Measure: Number; unit: Cases
Arm/Group | Study Ultrasound
Number analyzed (Participants) | 46
Cases | 29

ADVERSE EVENTS:
Time Frame: Participation in the proposed study did not pose any risks to the participants beyond what was expected from the standard of care stone management. Study PI monitored the study for any adverse events from the time of the study RBUS to day 42 post diagnostic CT. The timeframe in which data for adverse events was collected for this study was up to 45 days.
Arm/Group | Study Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT02577146/Prot_SAP_000.pdf